CLINICAL TRIAL: NCT05214079
Title: Determination of the Left Paratrachéal Force Required to Occlude the Esophageal Entrance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, MD, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Strenght_LPP
Record Dates: First submitted 2022-01-14; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Oesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 , Left paratracheal pressure (Active Comparator): 50 male
  Interventions: Device: Left paratracheal pressure
- 2, Left paratracheal pressure (Active Comparator): 50 female
  Interventions: Device: Left paratracheal pressure

INTERVENTIONS:
Device: Left paratracheal pressure — Applying Left Paratracheal pressure and testing its effectiveness using gastric tube . in addition , by using the dynamometer , the CP 50 is defined.

SUMMARY:
Determine the force required to occlude the esophagus with a left paratracheal pressure

ELIGIBILITY:
Inclusion Criteria:

* Physical status score 1 or 2
* No contre indication to Left Paratracheal pressure

Exclusion Criteria:

* Obese patients
* Physical status score 3, 4 or 5
* Contre indication to Left Paratracheal pressure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Necessary force of Left paratracheal pressure to occlude the esophagus in female versus male . an up and down method will define the CP 50 in each gender. A comparison between CP50 in both sex will define exactly our outcome | 24 hours